CLINICAL TRIAL: NCT00450190
Title: User Trial on the Use in Common Practice of a New Electronic Auto-injector of Saizen®, the E-Device (Electronic Device), in Children Treated by Recombinant Human Growth Hormone Over a Period of 2 Months
Brief Title: Saizen® E-Device User Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26443
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-09

CONDITIONS: Growth Disorders
Keywords: Growth disorders
MeSH Terms: conditions — Growth Disorders

ARMS (1):
- Saizen® E-Device (Experimental)
  Interventions: Device: Saizen® E-Device

INTERVENTIONS:
Device: Saizen® E-Device — Saizen® (recombinant human growth hormone [r-hGH]) injection 8 milligram (mg) per 137 milliliter (mL) will be administered using an electronic auto-injector (E-Device) subcutaneously (SC) in the evening as per local Summary of Product Characteristics (SmPC) for 60 days.

SUMMARY:
The aim of the study is to evaluate the E-Device performances and handling on the use in common practice, by collecting the impressions of patients, nurses and the investigator on the graphic interface, the instructions manual, the E-Device training and the material itself.

ELIGIBILITY:
Inclusion Criteria:

1. Patients naïve to, or experienced with, Saizen® with growth disorders in registered indications (GHD, Turner's Syndrome, Chronic Renal Failure, patient born Small Gestational Age [SGA] according to the local SmPC)
2. Written informed consent must be obtained from the parent(s)/legal guardian(s) at the beginning of the study. Children able to understand the trial should personally sign and date the written informed consent

Exclusion Criteria:

1. Known hypersensitivity to somatropin or any of the excipients
2. Epiphyseal fusion
3. Active neoplasia (either newly diagnosed or recurrent)
4. History of intracranial hypertension with papilledema
5. Diabetes mellitus or history of significant glucose intolerance as defined by a fasting blood glucose > 116 mg/dL
6. Severe congenital malformations
7. Severe psychomotor retardation
8. Known hepatic disease as defined by elevated liver enzymes or total bilirubin (x 2 N)
9. Current congestive heart failure, untreated hypertension, serious chronic oedema of any cause
10. Chronic infectious disease
11. Previous or ongoing treatment with sex steroid therapy such as estrogens and testosterone
12. Previous or ongoing treatment with any therapy that may directly influence growth, including GH, GHRF and long duration corticosteroids therapy
13. Proliferative or preproliferative diabetic retinopathy
14. Evidence of any progression or recurrence of an underlying intra-cranial space occupying lesion
15. Precocious puberty
16. Severe associated pathology affecting growth such as malnutrition, malabsorption or bone dysplasia
17. Concomitant corticoid treatment or levothyroxine treatment other than substitutive treatment, topical or inhaled treatment
18. Participation to any clinical study within the 30 days preceding study entry
19. Pregnancy

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02-28 (Actual); Primary Completion 2006-09-30 (Actual); Study Completion 2006-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Lipha Santé s.a.s., an affiliate of Merck KGaA, Darmstadt, Germany

REFERENCES:
- [Result] Tauber M, Payen C, Cartault A, Jouret B, Edouard T, Roger D. User trial of Easypod, an electronic autoinjector for growth hormone. Ann Endocrinol (Paris). 2008 Dec;69(6):511-6. doi: 10.1016/j.ando.2008.04.003. Epub 2008 Jun 26. PMID 18589398
- See also: Full FDA approved prescribing information can be found here — http://www.saizenus.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Saizen® E-Device: Saizen® (recombinant human growth hormone [r-hGH]) injection 8 milligram (mg) per 137 milliliter (mL) was administered using an electronic auto-injector (E-Device) subcutaneously (SC) in the evening as per local Summary of Product Characteristics (SmPC) for 60 days.
Period: Overall Study
Arm/Group | Saizen® E-Device
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Saizen® E-Device
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.30 (2.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Subjects' Overall Impression After Using E-Device
Description: Subjects' overall impression after using E-Device was measured on a scale ranging from 1 to 3, where 1 = bad, 2 = good, and 3 = very good. Number of subjects with response based on overall impression scale were presented.
Time Frame: 2 Weeks
Population: All subjects who were administered with at least 1 dose of study medication with E-Device.
Measure: Number; unit: subjects
Arm/Group | Saizen® E-Device
Number analyzed (Participants) | 20
subjects
  Bad | 0
  Good | 7
  Very Good | 13

2. Primary Outcome: Usefulness and Reliability of E-Device Functions
Description: Following functions were assessed: Display of remaining dose in cartridge, Display of last injection date and time, Automatic needle attachment, Audible and visual signals, Dose injected confirmation, Dose history, Customizable needle insertion speed, Customizable drug insertion speed, Customizable insertion depth, Teach me menu, On screen instructions, Customizable name and picture, Pre-programmed dose and Skin sensor. Usefulness and reliability of each of the E-Device functions was measured on a scale ranging from 1 to 3, where 1 = not useful, 2 = useful, and 3 = very useful. Number of subjects with response based on usefulness and reliability scale were presented.
Time Frame: 2 Weeks
Population: All subjects who were administered with at least 1 dose of study medication with E-Device.
Measure: Number; unit: subjects
Arm/Group | Saizen® E-Device
Number analyzed (Participants) | 20
subjects
  Display of remaining dose in cartridge: Not Useful | 0
  Display of remaining dose in cartridge: Useful | 8
  Display of remaining dose in cartridge:Very Useful | 12
  Display of last injection date/time: Not Useful | 3
  Display of last injection date/time: Useful | 11
  Display of last injection date/time: Very Useful | 6
  Automatic needle attachment: Not Useful | 0
  Automatic needle attachment: Useful | 9
  Automatic needle attachment: Very Useful | 11
  Audible and visual signals: Not Useful | 1
  Audible and visual signals: Useful | 9
  Audible and visual signals: Very Useful | 10
  Dose injected confirmation: Not Useful | 2
  Dose injected confirmation: Useful | 10
  Dose injected confirmation: Very Useful | 8
  Dose history: Not Useful | 5
  Dose history: Useful | 10
  Dose history: Very Useful | 5
  Customizable needle insertion speed: Not Useful | 2
  Customizable needle insertion speed: Useful | 9
  Customizable needle insertion speed: Very Useful | 9
  Customizable drug insertion speed: Not Useful | 1
  Customizable drug insertion speed: Useful | 11
  Customizable drug insertion speed: Very Useful | 8
  Customizable insertion depth: Not Useful | 1
  Customizable insertion depth: Useful | 9
  Customizable insertion depth: Very Useful | 10
  Teach me menu: Not Useful | 8
  Teach me menu: Useful | 7
  Teach me menu: Very Useful | 5
  On screen instructions: Not Useful | 0
  On screen instructions: Useful | 6
  On screen instructions: Very Useful | 14
  Customizable name and picture: Not Useful | 13
  Customizable name and picture: Useful | 7
  Customizable name and picture: Very Useful | 0
  Pre-programmed dose: Not Useful | 0
  Pre-programmed dose: Useful | 6
  Pre-programmed dose: Very Useful | 14
  Skin sensor: Not Useful | 2
  Skin sensor: Useful | 8
  Skin sensor: Very Useful | 10

3. Secondary Outcome: Subjects' Feedback Immediately After Initial Training During Inclusion Visit
Description: Subjects' feedback immediately after initial training on the handling and use of E-Device was assessed on scale ranging from 1 to 3, where 1 = difficult, 2 = easy, and 3 = very easy. Subjects were provided training on the following aspects: Cartridge loading, Needle attachment, Needle detachment, Injection process, Navigation in the menu, and Handling of the device. Number of subjects with response based on their feedback were presented.
Time Frame: Inclusion visit (Day 1)
Population: All subjects who were administered with at least 1 dose of study medication with E-Device.
Measure: Number; unit: subjects
Arm/Group | Saizen® E-Device
Number analyzed (Participants) | 20
subjects
  Cartridge loading: Difficult | 1
  Cartridge loading: Easy | 17
  Cartridge loading: Very Easy | 2
  Needle attachment: Difficult | 2
  Needle attachment: Easy | 15
  Needle attachment: Very Easy | 3
  Needle detachment: Difficult | 7
  Needle detachment: Easy | 12
  Needle detachment: Very Easy | 1
  Injection process: Difficult | 1
  Injection process: Easy | 16
  Injection process: Very Easy | 1
  Injection process: Missing data | 2
  Navigation in the menu: Difficult | 2
  Navigation in the menu: Easy | 17
  Navigation in the menu: Very Easy | 1
  Handling of the device: Difficult | 1
  Handling of the device: Easy | 15
  Handling of the device: Very Easy | 0
  Handling of the device: Missing data | 4

4. Secondary Outcome: Nurse/Physician's Feedback After E-Device Set up During Inclusion Visit
Description: Nurse/physician's feedback was assessed for E-Device setting up and Dose programming on inclusion visit using a scale ranging from 1 to 3, where 1 = difficult, 2 = easy, and 3 = very easy. Nurse/Physician's response for the number of subjects were presented.
Time Frame: Inclusion visit (Day 1)
Population: All included subjects were analyzed who used at least 1 dose of study medication with E-Device.
Measure: Number; unit: subjects
Arm/Group | Saizen® E-Device
Number analyzed (Participants) | 20
subjects
  Device setting up: Difficult | 1
  Device setting up: Easy | 19
  Device setting up: Very Easy | 0
  Dose programming: Difficult | 0
  Dose programming: Easy | 19
  Dose programming: Very Easy | 0
  Dose programming: Missing data | 1

5. Secondary Outcome: Number of Subjects With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A Serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect, AEs leading to discontinuation and AEs leading to death.
Time Frame: Day 1 up to Day 90
Population: All subjects who were administered with at least 1 dose of study medication with E-Device.
Measure: Number; unit: subjects
Arm/Group | Saizen® E-Device
Number analyzed (Participants) | 20
subjects
  AEs | 0
  SAEs | 0

ADVERSE EVENTS:
Arm/Group | Saizen® E-Device
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other